CLINICAL TRIAL: NCT05648812
Title: Contrast Enhanced Ultrasound and Elastography of the Neonatal Brain
Brief Title: Neonatal Brain Ultrasound With CEUS and Elastography
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Tiina Laurikainen, Principal Investigator, Turku University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TL16102021
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Hypoxic Ischemic Encephalopathy; Neonatal Stroke; Neonatal Encephalopathy, Unspecified
MeSH Terms: interventions — Sulfur Hexafluoride; contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Term neonates (Active Comparator): Diagnostic Test: Brain ultrasound, brain contrast enhanced ultrasound, brain ultrasound elastography, cardiac ultrasound To study brain perfusion with brain ultrasound, contrast enhanced ultrasound of the brain and ultrasound-guided shear-wave elastography Drug: Sulfur Hexafluoride To evaluate brain perfusion in infants with no suspected brain pathology using CEUS. Later, different patient groups could be compared to infants with no suspected brain pathology.
  Other Names:
  • SonoVue
  Interventions: Diagnostic Test: Brain contrast enhanced ultrasound, brain ultrasound elastography; Drug: Sulfur Hexafluoride
- Neonatal asphyxia (Experimental): Diagnostic Test: Brain ultrasound, brain contrast enhanced ultrasound, brain ultrasound elastography To study brain perfusion with brain ultrasound, contrast enhanced ultrasound of the brain and ultrasound-guided shear-wave elastography Drug: Sulfur Hexafluoride To evaluate brain perfusion in neonates after birth asphyxia
  Other Names:
  • SonoVue
  Interventions: Diagnostic Test: Brain contrast enhanced ultrasound, brain ultrasound elastography; Drug: Sulfur Hexafluoride
- Neonatal stroke (Experimental): Diagnostic Test: Brain contrast enhanced ultrasound, brain ultrasound elastography To study brain perfusion with brain ultrasound, contrast enhanced ultrasound of the brain and ultrasound-guided shear-wave elastography Drug: Sulfur Hexafluoride To evaluate brain perfusion after neonatal stroke
  Other Names:
  • SonoVue
  Interventions: Diagnostic Test: Brain contrast enhanced ultrasound, brain ultrasound elastography; Drug: Sulfur Hexafluoride
- Other neonatal brain pathologies (Experimental): Diagnostic Test: Brain ultrasound, brain contrast enhanced ultrasound, brain ultrasound elastography To study brain perfusion with brain ultrasound, contrast enhanced ultrasound of the brain and ultrasound-guided shear-wave elastography Drug: Sulfur Hexafluoride To evaluate brain perfusion in infants with other type (no asphyxia, stroke or preterm birth related) of brain pathology, like hydrocephalus, hemorrhage or central nervous system infection
  Other Names:
  • SonoVue
  Interventions: Diagnostic Test: Brain contrast enhanced ultrasound, brain ultrasound elastography; Drug: Sulfur Hexafluoride

INTERVENTIONS:
Diagnostic Test: Brain contrast enhanced ultrasound, brain ultrasound elastography — To study brain perfusion with brain ultrasound, contrast enhanced ultrasound of the brain and ultrasound-guided shear-wave elastography
Drug: Sulfur Hexafluoride — To evaluate the differences in brain perfusion studied by CEUS, comparing different patient groups and babies with no suspected brain pathology
  Other Names: SonoVue

SUMMARY:
The aim of our study is to investigate changes of brain perfusion and elasticity in neonates during the time that a neonate is adapting to live outside the womb and during diseases that are suspected to affect neonatal brain perfusion. We use contrast enhanced ultrasound (sulphur hexafluoride) and ultrasound-assisted elastography to evaluate the state of brain perfusion. We will study neonates recruited from the Neonatal Units of Turku University Hospital.

DETAILED DESCRIPTION:
SonoVue (sulphur hexafluoride) is a contrast agent composed of micro bubbles. It increases echogenicity of the ultrasound thus enhancing the visualisation of vessels and giving better insights into tissue perfusion. The use of sulphur hexafluoride has been approved by FDA and it has been in off-label use in Europe for years. SonoVue is thought to be especially useful for children, because it can enhance the diagnostic capabilities of ultrasound and the examination can be performed without radiation or sedation.

Elastography is a method to investigate the elasticity of a tissue by tracking the shear waves generated by the ultrasound beam. Also this method has been used in Europe and America for years.

The aim of our study is to examine cerebral hemodynamics in neonates using ultrasound of the brain, contrast enhanced ultrasound (CEUS) and ultrasound-guided shear-wave elastography (US-SWE). We aim to recruit four groups of infants: those with no suspected diseases affecting brain perfusion on the first days after birth and infants with either asphyctic injury, stroke or other diseases affecting central nervous system. Total recruitment for different groups is 100 infants in total, during this first study phase. The recruitment period will be up to seven years if needed.

The injections of SonoVue will be administered through pre-existing venous cannulas. The first examination after brain injury will be done as soon as the parental consent has been given. The ultrasound examination altogether is estimated to take about 20 minutes per day. Safety monitoring period is conducted after the injection. The studies will be repeated 0-4 times according to the approval of the caretakers of the child and the disease the child is affected by. CEUS data will be analysed with proper software. US-SWE will be measured repeatedly on both brain hemispheres and on different areas to validate the measurements.

ELIGIBILITY:
Inclusion Criteria:

* Babies less than 7 months treated at the neonatal units of Turku University hospital

Exclusion Criteria:

* Pre-known genetic disease
* Difficult congenital malformations that need surgical treatment
* Central nervous system tumors
* Weight less than 2,5 kg during examination
* Medical history of SonoVue hypersensitivity
* Uncontrolled systemic hypertension
* Systolic pulmonary artery pressure > 90 mmHg
* Unstable cardiovascular state

Ages: 1 Minute to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Repeated qualitative and quantitative assessment of neonatal brain perfusion using contrast-enhanced ultrasound of the brain | 20 days
  Visual assessment of contrast enhancement on both brain hemispheres. Quantitative analysis of proper ultrasound parameters, such as wash-in and wash-out curves, during the adaptive period and during different brain pathologies and their treatment.

SECONDARY OUTCOMES:
Repeated qualitative assessment of neonatal brain elasticity using ultrasound-guided shear wave elastography | 20 days
  Quantitative analysis of repeated US-SWE measurements on both hemispheres and areas of interest estimated by brain ultrasound and CEUS
Comparing the brain perfusion in neonates with no diseases affecting brain perfusion and neonates with different brain pathologies | 20 days
  Quantitative analysis of proper contrast-enhanced ultrasound parameters, such as wash-in and wash-out curves, in neonates with normal brain perfusion compared to neonates with different brain pathologies.

CONTACTS AND LOCATIONS:
Overall Officials: Tiina Laurikainen, Principal Investigator — Turku University Hospital; Riitta Parkkola, Study Director — Turku University Hospital; Vilhelmiina Parikka, Study Chair — Turku University Hospital; Jussi Hirvonen, Study Chair — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Southwestern Finland, Finland

IPD SHARING:
Plan to Share IPD: No